CLINICAL TRIAL: NCT07077811
Title: The Safety and Efficacy of Pulsed Field Ablation for Patients With Persistent Atrial Fibrillation Comorbid With HFpEF: a Prospective, Multicenter Cohort Study
Brief Title: The Safety and Efficacy of Pulsed Field Ablation for Patients With Persistent Atrial Fibrillation Comorbid With HFpEF.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-K119-01
Record Dates: First submitted 2025-06-15; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Heart Failure; Atrial Fibrillation (AF); HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: Persistent Atrial Fibrillation; Heart Failure with Preserved Ejection Fraction; Pulsed field ablation
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical group (Experimental): Medtronic Pulse Select pulsed field ablation Group
  Interventions: Procedure: pulsed field ablation
- Drug group (Active Comparator): Group treated with class I or class III antiarrhythmic drugs
  Interventions: Drug: antiarrhythmic drug

INTERVENTIONS:
Procedure: pulsed field ablation — Medtronic Pulse Select pulsed field ablation
  Arms: Surgical group
Drug: antiarrhythmic drug — treated with class I or class III antiarrhythmic drugs
  Arms: Drug group

SUMMARY:
The goal of this clinical trial is to evaluate the the mid- and long-term clinical efficacy and safety of pulsed field catheter ablation for patients with persistent atrial fibrillation and HFpEF. The main questions it aims to answer are:

* What are the differences between the effects of pulsed field ablation and drug therapy?
* Which risk factors affecting the outcome of atrial fibrillation ablation, postoperative recurrence, and improvement of cardiac function? Researchers will compare pulsed field ablation to drug therapy to provide some theoretical basis and clinical evidence for the treatment strategy of patients with atrial fibrillation and HFpEF.

This study selected patients with persistent AF and HFpEF and divided them into a drug group (treated with class I or class III antiarrhythmic drugs) and a surgical group (Medtronic Pulse Select pulsed field ablation).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common arrhythmias in clinical practice. It is a supraventricular tachyarrhythmia characterized by rapid and disordered atrial electrical activity, with a high disability and mortality rate. Atrial fibrillation not only significantly reduces the patient's cardiac output, leading to heart failure；It will also increase the risk of left atrial mural thrombus formation, leading to peripheral arterial embolism, especially stroke. AF is currently the most common arrhythmia in patients with heart failure (HF). Studies have shown that atrial fibrillation is more common in patients with ejection fraction preserving heart failure (HFpEF). During the course of HFpEF, atrial dysfunction caused by atrial fibrillation may cause functional mitral regurgitation, further affecting ventricular systolic and diastolic function and accelerating the progression of heart failure. Patients with atrial fibrillation and heart failure have severe symptoms, poor prognosis, and increased hospitalization rates.

The goal of treating atrial fibrillation combined with heart failure is to alleviate patient symptoms and improve survival rate. The treatment strategies for atrial fibrillation mainly include standardized anticoagulation therapy and catheter ablation. Catheter ablation includes catheter ablation under high-power X-ray guidance, radiofrequency ablation guided by a three-dimensional mapping system, radiofrequency ablation guided by intracardiac ultrasound, high-power short-term radiofrequency ablation, cryoballoon ablation, pulsed field ablation, left atrial appendage occlusion, and "one-stop treatment for atrial fibrillation". Studies have reported that for patients with heart failure and atrial fibrillation, compared with drug treatment, radiofrequency catheter ablation significantly reduces all-cause mortality and heart failure hospitalization rate, and significantly improves cardiac function classification.

Pulsed field ablation (PFA) is an emerging ablative energy. The basis for the damage effect of ablation is the voltage difference between the inside and outside of the membrane formed by the high-voltage electric field. This is electric field-dependent, does not generate heat locally, and has strong penetration ability. Under the action of high-voltage electric fields, the damage threshold of different tissues is different. The damage is selective to a certain extent, and it is safer for fragile adjacent tissues such as blood vessels, esophagus, and nerves. Currently, other energy forms used for ablation are not selective for this tissue type. In the global key study, the incidence of unsafe events for the product submitted this time was 0.7%, and no complications such as left atrial-esophageal fistula, pulmonary vein stenosis, myocardial infarction, phrenic nerve palsy, and coronary spasm occurred. The extremely low incidence of unsafe events demonstrates the excellent safety of the product. Compared with existing technologies, the efficiency of PFA energy may also be improved. PFA delivery is completed in a few milliseconds, which may reduce isolation time and the entire operation time. By reducing the total operation time, the anesthesia time and the time the patient and doctor are exposed to radiation are reduced, which greatly improves the efficiency of the operation. The PulseSelect™ pulsed field ablation system is a ring electrode with a central support. Compared with a point-shaped radiofrequency catheter, it isolates the pulmonary veins by ablating a whole circle of 9 electrodes at the same time, further improving the efficiency of the operation. Due to the uniqueness and safety of its energy, it can significantly reduce postoperative complications and hospitalization time, shorten the patient's recovery period, and reduce the need for secondary treatment, thereby effectively reducing the patient's medical costs and economic burden. The results of the Pulsed AF study also showed that at 6 and 12 months after surgery, the overall quality of life of patients (AFEQT and EQ-5D) increased by 5 points and 0.03 points respectively compared with the baseline level, and the results were statistically significant. It can be seen that PFA reduces the overall medical resource investment by reducing the re-ablation rate and cardiovascular events.

In summary, patients with persistent atrial fibrillation and HFpEF have a poor prognosis and lack effective treatment. This study is dedicated to treating patients with persistent atrial fibrillation and HFpEF with pulsed field catheter ablation, and will follow up for 12 months to evaluate the effectiveness and safety of pulsed field catheter ablation for these patients. It is hoped that this study will bring new hope to patients with atrial fibrillation and HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;
* Patients with persistent atrial fibrillation;
* According to the 2021 European Society of Cardiology (ESC) guidelines for heart failure, heart failure with preserved ejection fraction (HFpEF) is defined as patients with preserved or slightly reduced left ventricular ejection fraction (LVEF) but with diastolic dysfunction. The diagnostic criteria for HFpEF include: symptoms and signs of heart failure; LVEF≥50%; and objective evidence of cardiac structural and functional abnormalities consistent with left ventricular diastolic dysfunction or increased left ventricular filling pressure. These can be verified by imaging examinations such as echocardiography and biomarkers such as B-type natriuretic peptide or NT-proBNP. The thresholds for B-type natriuretic peptide or NT-proBNP are: BNP≥35 pg/mL or NT-proBNP ≥125 pg/mL for patients with sinus rhythm; BNP≥105 pg/mL or NT-proBNP ≥365 pg/mL for patients with atrial fibrillation.
* Agree to participate in this study and sign the informed consent form. Have clinical compliance to complete the postoperative follow-up required by the protocol.

Exclusion Criteria:

* Patients with persistent atrial fibrillation lasting for more than 3 years;
* Patients who had used class I or class III antiarrhythmic drugs, but the use of the above drugs for less than 7 days to convert atrial fibrillation was allowed;
* Previous left atrial ablation or surgery (including left atrial appendage occlusion);
* Left atrial diameter > 50 mm;
* Previous pulmonary vein stenting;
* Previous pulmonary vein stenosis;
* Presence of any heart valve prosthesis;
* Any cardiac surgery, myocardial infarction, percutaneous coronary intervention (PCI)/percutaneous transluminal coronary angioplasty (PTCA) or coronary artery stenting within three months before signing the informed consent;
* Unstable angina or severe coronary artery stenosis;
* Primary pulmonary hypertension;
* Rheumatic heart disease;
* Thrombocytosis, thrombocytopenia;
* Any disease that prohibits long-term anticoagulation;
* Active systemic infection;
* Atrial fibrillation caused by reversible causes, such as hyperthyroidism;
* Women known to be pregnant or breastfeeding;
* Life expectancy of less than one year;
* Patients with intracardiac thrombus;
* Patients with known drug or alcohol addiction;
* Patients who are unwilling or unable to fully comply with the study protocol and complete follow-up;
* Patients with malignant tumors;
* Participating in other clinical trials that may interfere with the results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life at 12 months as measured by the Atrial Fibrillation Quality of Life Survey (AFEQT). | 12 months
  Improvement in quality of life from baseline to 12 months after pulsed field ablation procedure or AAD as measured by the Atrial Fibrillation Quality of Life Survey (AFEQT), with values ranging from 20 - 140 (higher scores mean worse outcomes).

SECONDARY OUTCOMES:
The rate of atrial fibrillation-free recurrence | 12 months after surgery
  The rate of atrial fibrillation-free recurrence during clinical follow-up within 12 months after surgery, that is, the success rate of pulsed field therapy for AF (including atrial tachycardia (AT) lasting more than 30 seconds, atrial flutter (AFL), and AF endpoint events;
Complications and adverse events | perioperative period
  Complications and adverse events during the pulsed field ablation surgery and during the postoperative follow-up, including readmission, cardiovascular events, cardiovascular death, all-cause death, and also including serious adverse events related to the surgery.
Readmission Rate | 3 months after surgery
  Rehospitalization due to heart failure or recurrence of atrial fibrillation 3 months after surgery
The incidence of AT/AF/AFL events | 3 months after surgery
  The incidence of AT/AF/AFL events 3 months later;
Improvement of cardiac function | 6 and 12 months after surgery
  echocardiogram E/e'

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT07077811/Prot_000.pdf